CLINICAL TRIAL: NCT00292916
Title: Effect of Whole Body Vibration on Bone and Fall Related Parameters - the Erlangen Longitudinal Vibration Study (ELVIS)
Brief Title: Effect of Whole Body Vibration on Bone and Fall Related Parameters
Status: Terminated | Phase: Phase 3 | Type: Interventional
Sponsor: University of Erlangen-Nürnberg Medical School (Other)
Collaborators: Institute of Biometrie and Medical Statistics (Unknown); Netzwerk-Knochengesundheit (Unknown); Siemens-Betriebskrankenkasse (Industry)
Responsible Party: Principal Investigator, Wolfgang Kemmler, Principal Investigator, University of Erlangen-Nürnberg Medical School
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: D-ER-OFZ-200501-Vib
Record Dates: First submitted 2006-02-15; First posted 2006-02-16 (Estimated); Last update posted 2015-05-28 (Estimated); Status verified 2015-05

CONDITIONS: Atrophy
Keywords: whole body vibration; exercise; elderly woman; Bone Mineral Density; falls; higher age
MeSH Terms: conditions — Atrophy; Motor Activity | interventions — Resistance Training; Health

INTERVENTIONS:
Behavioral: whole body vibration
Behavioral: resistance exercise
Behavioral: "wellness"

SUMMARY:
The effect of whole body vibration (WBV) on bone strength and fall frequency in older adults is still vague. Although there is some evidence that WBV may impact Bone Mineral Density in very frail elderly, there is a lack of data concerning the effect of WBV in community-living elderly woman. We hypothesize that WBV significantly affects bone parameters as assessed by DXA, QCT, US and bone markers with parallel positive changes of fall related risk factors (power, strength, balance, and reaction time). We further hypothesize that the effects of WBV were superior to conventional resistance exercise.

ELIGIBILITY:
Inclusion Criteria:

* community living elderly females >/=65 years
* live expectation > 2 years

Exclusion Criteria:

* secondary osteoporosis
* CVD-events including stroke
* participation in other studies
* medication and illness affecting bone metabolism within the last 2 years
* medication with impact on falls
* low physical performance (<50 Watt during ergometry)
* excessive alcohol-intake

Min Age: 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 150
Dates: Start 2006-01; Study Completion 2007-07 (Actual)

PRIMARY OUTCOMES:
BMD after 6, 12 and 18 months
strength
power

SECONDARY OUTCOMES:
balance
bone markers

CONTACTS AND LOCATIONS:
Overall Officials: Willi A Kalender, PhD, Study Chair — University of Erlangen-Nürnberg Medical School
Locations (1):
- Institute of Medical Physics, Erlangen, Germany

REFERENCES:
- [Background] Kemmler W, Engelke K, Baumann H, Beeskow C, von Stengel S, Weineck J, Kalender WA. Bone status in elite male runners. Eur J Appl Physiol. 2006 Jan;96(1):78-85. doi: 10.1007/s00421-005-0060-1. Epub 2005 Oct 26. PMID 16307280
- [Background] Engelke K, Kemmler W, Lauber D, Beeskow C, Pintag R, Kalender WA. Exercise maintains bone density at spine and hip EFOPS: a 3-year longitudinal study in early postmenopausal women. Osteoporos Int. 2006 Jan;17(1):133-42. doi: 10.1007/s00198-005-1938-9. Epub 2005 Aug 12. PMID 16096715
- [Background] Stengel SV, Kemmler W, Pintag R, Beeskow C, Weineck J, Lauber D, Kalender WA, Engelke K. Power training is more effective than strength training for maintaining bone mineral density in postmenopausal women. J Appl Physiol (1985). 2005 Jul;99(1):181-8. doi: 10.1152/japplphysiol.01260.2004. Epub 2005 Mar 3. PMID 15746294
- [Background] Kemmler W, Weineck J, Kalender WA, Engelke K. The effect of habitual physical activity, non-athletic exercise, muscle strength, and VO2max on bone mineral density is rather low in early postmenopausal osteopenic women. J Musculoskelet Neuronal Interact. 2004 Sep;4(3):325-34. PMID 15615501
- [Derived] Von Stengel S, Kemmler W, Bebenek M, Engelke K, Kalender WA. Effects of whole-body vibration training on different devices on bone mineral density. Med Sci Sports Exerc. 2011 Jun;43(6):1071-9. doi: 10.1249/MSS.0b013e318202f3d3. PMID 20980923